CLINICAL TRIAL: NCT07032480
Title: Association Between Sleep Disorders, Neck Pain, and Depression in Young Adults: A Cross-Sectional Study
Brief Title: Association Between Sleep Disorders, Neck Pain, and Depression
Status: Recruiting | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, ESRA PEHLIVAN, Principal Investigator, Saglik Bilimleri Universitesi
Other Study IDs: Sleep&Neck&Depression
Record Dates: First submitted 2025-06-14; First posted 2025-06-24 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Health Risk Behaviors
MeSH Terms: conditions — Health Risk Behaviors

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy Sleep Group: Participants who scored 0-5 on the Pittsburgh Sleep Quality Index (PSQI), indicating good sleep quality.
  Interventions: Behavioral: Survey-Based Assessment
- Poor Sleep Group: Participants who scored between 6-10 on the PSQI, indicating impaired sleep quality.
  Interventions: Behavioral: Survey-Based Assessment
- Chronic Sleep Disorder Group: Participants who scored above 10 on the PSQI, indicating persistent and clinically relevant sleep disturbances.
  Interventions: Behavioral: Survey-Based Assessment

INTERVENTIONS:
Behavioral: Survey-Based Assessment — Participants completed standardized questionnaires including the Beck Depression Inventory (BDI), Pittsburgh Sleep Quality Index (PSQI), and Neck Disability Index (NDI) to evaluate psychological and functional outcomes associated with sleep quality. No experimental intervention was administered.

SUMMARY:
This cross-sectional observational study investigates the association between sleep quality, neck pain-related disability, and depression symptoms in young adults aged 18-28. The research reveals that poor sleep quality is significantly associated with higher depression scores and increased neck disability, emphasizing the need for integrative approaches targeting sleep quality to improve mental and musculoskeletal health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-28
* No history of physical or psychological illness
* Able to provide informed consent
* Voluntarily agreed to participate

Exclusion Criteria:

* History of chronic illness or psychiatric disorder
* Communication difficulties

Ages: 18 Years to 28 Years | Sex: All
Age Groups: Adult
Study Population: Healthy young adults aged 18-28 residing in Istanbul, Turkey. Participants were recruited via university student pools and personal networks of the researchers.
Sampling Method: Non-Probability Sample
Enrollment: 265 (Estimated)
Dates: Start 2025-06-26 (Actual); Primary Completion 2026-06-22 (Estimated); Study Completion 2026-06-22 (Estimated)

PRIMARY OUTCOMES:
Sleep Quality as Measured by the Pittsburgh Sleep Quality Index (PSQI) | Single assessment at baseline
  The PSQI is a validated self-report instrument that evaluates sleep quality and disturbances over a 1-month period. It includes 7 subscales: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. Each component is scored from 0 (no difficulty) to 3 (severe difficulty), resulting in a global score from 0 to 21.

SECONDARY OUTCOMES:
Functional Neck Disability as Measured by the Neck Disability Index (NDI) | Single assessment at baseline
  The NDI is a 10-item questionnaire that assesses how neck pain affects daily activities such as personal care, lifting, reading, concentration, work, driving, sleeping, and recreation. Each item is scored from 0 to 5, for a total possible score of 0 to 50.
Depression Severity as Measured by the Beck Depression Inventory (BDI) | Single assessment at baseline
  The BDI is a 21-item self-report questionnaire assessing depressive symptoms in individuals. Each item is rated on a 4-point scale (0 to 3), with a total possible score ranging from 0 to 63. Higher scores indicate more severe depressive symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Saglik Bilimleri Universitesi, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided